CLINICAL TRIAL: NCT05199376
Title: Evaluation of Percutaneous Cryotherapy in the Treatment of Plexiform Neurofibromas and Unresectable Neurofibromas in Neurofibromatosis Type 1 (NF1)
Brief Title: Evaluation of Percutaneous Cryotherapy in the Treatment of Plexiform Neurofibromas and Unresectable Neurofibromas in Neurofibromatosis Type 1
Acronym: CryoNF1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET21-198
Record Dates: First submitted 2021-12-21; First posted 2022-01-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Neurofibroma; Neurofibroma, Plexiform
MeSH Terms: conditions — Neurofibroma; Neurofibroma, Plexiform | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous cryotherapy (Experimental): Cryoablation of the tumor
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Cryotherapy — The cryotherapy treatment lasts approximately 30 minutes during which two 10-minute freezing cycles are performed, separated by a reheating phase. During the freezing phases, the temperature is lowered below -40°C in the ablation zone, a temperature that is lethal for the cells.

SUMMARY:
Neurofibromatosis type 1 (NF1) is an autosomal dominant disease affecting chromosome 17. It is manifested by a neurogenic tumor proliferation that forms cutaneous, subcutaneous or deep neurofibromas.

Neurofibromas can cause functional discomfort, neurogenic pain that is difficult to treat, and severe cosmetic disorders.

Treatment is essentially surgical. It is sometimes a heavy invasive surgery with complicated postoperative follow-up and significant scarring on the aesthetic level. Currently, no systemic treatment has proven its effectiveness in this pathology.

Percutaneous cryotherapy is a cold thermoablation procedure using fine 17 G needles introduced into the lesion after targeting by imaging. This technique is used in the treatment of soft tissue tumors and desmoid tumors.

The treatment of neurofibromas with percutaneous cryotherapy is not well known. Encouraging results (unpublished) have been observed in patients with NF1 treated with cryotherapy at the Léon Bérard Center. The beneficial effect was observed in terms of quality of life (in particular, pain) as well as a decrease in tumor size.

On the basis of this first experience, it appears important to corroborate these preliminary results by a prospective study allowing the use of this technique to treat patients with unresectable or resectable neurofibromas but with mutilating surgery in a NF1 context.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Patient with neurofibromatosis type 1 according to NIH criteria ;
* Patient with a benign neurofibromatous lesion that is painful and/or generates functional discomfort and is unresectable or with unacceptable scarring ;
* Neutrophils > 1 G/l in the 14 days prior to inclusion;
* Adequate coagulation test with normals values (as judged by the investigator);
* Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment
* Covered by a medical insurance;

Exclusion Criteria:

* Patient treated with concomitant chemotherapy and/or targeted therapies ;
* Any contraindication to a percutaneous cryotherapy procedure, including the need for ice formation within 1 cm of the spinal cord, brain or other critical nerve structures, bowel or bladder (unless active or passive thermal protective maneuvers are performed);
* Patient with malignant neurofibroma or MPNST ; CT scan without abnormality and if tumor presents a max SUV T/F>1.5 ratio, targeted biopsy is required to confirm benign or malignant histology.
* Patient with neurofibroma in areas at risk for neurological sequelae;
* Patient with cold urticaria with history of angioedema;
* Any cognitive impairment or condition that may limit the use of numerical scales and quality of life questionnaires;
* Patient for whom follow-up does not seem feasible even in the short term;
* Participation in another clinical trial that may interfere with the evaluation of the primary endpoint;
* Patient under tutorshio, curatorship or deprived of liberty;
* Pregnant or breast-feeding woman;
* Any contraindication to the performance of an MRI
* Patient with dysplastic neurofibroma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2027-02-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of percutaneous cryotherapy on physical health-related quality of life (in patients with inoperable (or operable with mutilating surgery) neurofibroma. | 12 months after cryotherapy
  Rate of patients with clinically significant improvement in physical health-related quality of life.
  A patient will be considered successful if an increase of at least 3 points on the global physical score from the SF-36 questionnaire is observed at least once between baseline and 12 months after cryotherapy.

SECONDARY OUTCOMES:
To assess each quality of life dimension of the Short Form-36 (SF-36) questionnaire; | At baseline, at Month1 post cryotherapy ; Month 3 post cryotherapy; Month 6 post cryotherapy, Month 9 post cryotherapy, Month 12 post cryotherapy, Month 18 post cryotherapy and Month 24 post post cryotherapy ;
  The score for each dimension, the mental global score and the physical global score from the SF-36 questionnaire
To evaluate the tumor response | Month 3, Month 6, Month 9, Month 12, Month 18 , and Month 24 after cryotherapy
  Local control rate using REiNS and RECIST 1.1 criteria
To evaluate the functional discomfort | At baseline, Month 1; Month 3; Month 6, Month 9, Month12, Month18 and Month 24 post cryotherapy
  Functional discomfort assessed by a Likert scale
To evaluate the patients' pain | At baseline, Month 1; Month 3; Month 6, Month 9, Month 12, Month 18 and Month 24 post cryotherapy
  Pain assessed by the Brief Pain Inventory-Short Form (BPI-SF) questionnaire
To evaluate the safety of percutaneous cryotherapy | From cryotherapy to 24 months after cryotherapy
  Tolerance of cryotherapy treatment assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
To evaluate patients' satisfaction | At Month 12 post-cryotherapy;
  Patient satisfaction with their first cryotherapy treatment assessed by a Likert scale
To evaluate patients self-esteem | at baseline, Month 1; Month 3; Month 6, Month 9, Month12, Month 18 and Month 24 post-cryotherapy
  Self-esteem assessed by a questionnaire consisting of items evaluated on a Likert scale
To evaluate the need for multiple percutaneous cryotherapy procedures in case of incomplete response on the target lesion; | From cryotherapy to 24 months after cryotherapy
  Rate of patients for whom at least one additional percutaneous cryotherapy procedure is required
To evaluate operating room occupancy time. | At Day 0
  Median operating room occupancy time calculated as the difference between operating room exit time and operating room entry time.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Leon Berard, Lyon, France

IPD SHARING:
Plan to Share IPD: No